CLINICAL TRIAL: NCT01734057
Title: A Multicentre Investigation of Recombinant Human Thrombopoietin (rhTPO) Combining Rituximab Versus High-dose Dexamethasone for Initial Treatment of Primary Immune Thrombocytopenia (ITP)
Brief Title: Recombinant Human Thrombopoietin (rhTPO) Combining Rituximab Versus High-dose Dexamethasone for Initial Treatment of Primary Immune Thrombocytopenia (ITP)
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: No eligible patient was enrolled.
Sponsor: Shandong University (Other)
Collaborators: The Affiliated Hospital of the Chinese Academy of Military Medical Sciences (Other); Anhui Medical University (Other); The First Affiliated Hospital of Dalian Medical University (Other); Shandong Provincial Hospital (Other Government); Shenzhen Second People's Hospital (Other); China Medical University, China (Other); Zhejiang Provincial Hospital of TCM (Other)
Responsible Party: Principal Investigator, Ming Hou, Professor and Director, Shandong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ITP-008
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2012-11

CONDITIONS: Purpura; Idiopathic Thrombocytopenic Purpura
Keywords: Recombinant Human Thrombopoietin; rhTPO; Rituximab; Dexamethasone
MeSH Terms: conditions — Purpura; Purpura, Thrombocytopenic, Idiopathic | interventions — Thrombopoietin; Rituximab; Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- combinant treatment group (Experimental): 120 enrolled patients are randomly picked up to take Rituximab in combination with rhTPO at the indicated dose.
  Interventions: Drug: recombinant human thrombopoietin (rhTPO); rituximab
- single treatment group (Active Comparator): 120 enrolled patients are randomly picked up to take dexamethasone at the indicated dose.
  Interventions: Drug: Dexamethasone

INTERVENTIONS:
Drug: recombinant human thrombopoietin (rhTPO); rituximab — patients in recombination treatment group take Rituximab( intravenously ,100 mg weekly for 4 consecutive weeks); in combination with rhTPO( subcutaneously , 300U/kg for 14 consecutive days,followed by flexible treating dosage so as to keep the platelet count above 50×10^9/L until the 28th day)
  Other Names: Recombinant Human Thrombopoietin; Recombinant Human TPO; rhTPO combine with Rituximab; Recombinant Human Thrombopoietin combine with Rituximab; Recombinant Human TPO combine with Rituximab
  Arms: combinant treatment group
Drug: Dexamethasone — Patients in single treatment group take dexamethasone intravenously at 40 mg daily for 4 consecutive days.
  Arms: single treatment group

SUMMARY:
The project was undertaking by Qilu Hospital of Shandong University and other 13 well-known hospitals in China. In order to report the efficacy and safety of Recombinant Human thrombopoietin combining with Rituximab for the treatment of adults with primary immune thrombocytopenia (ITP), compared to conventional high-dose dexamethasone therapy.

DETAILED DESCRIPTION:
The investigators are undertaking a parallel group, multicentre, randomised controlled trial of 240 primary ITP adult patients from 14 medical centers in China. One part of the participants are randomly selected to receive recombinant human thrombopoietin (given subcutaneously at a dose of 300Units/kgfor 14 consecutive days, following with a flexible dosage depending on platelet count until the 28th day), combining with rituximab (given intravenously at a dose of 100 mg weekly for 4 weeks, i.e. Day 1, 8, 15, 22; the others are selected to receive high-dose of dexamethasone treatment (given intravenously at a dose of 40 mg daily for 4 days). Platelet count was evaluated before and after treatment,in order to report the conversion ratio of primary ITP to chronic ITP.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for immune thrombocytopenia.
2. Untreated hospitalized patients, may be male or female, between the ages of 18 ~ 80 years.
3. To show a platelet count < 30×10^9/L, and with bleeding manifestations.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Willing and able to sign written informed consent

Exclusion Criteria:

1. Received chemotherapy or anticoagulants or other drugs affecting the platelet counts within 3 months before the screening visit.
2. Received high-dose steroids or intravenous immunoglobulin transfusion(IVIG) in the 3 weeks prior to the start of the study.
3. Current HIV infection or hepatitis B virus or hepatitis C virus infections.
4. Severe medical condition (lung, hepatic or renal disorder) other than ITP. Unstable or uncontrolled disease or condition related to or impacting cardiac function (e.g., unstable angina, congestive heart failure, uncontrolled hypertension or cardiac arrhythmia)
5. Female patients who are nursing or pregnant, who may be pregnant, or who contemplate pregnancy during the study period.
6. Have a known diagnosis of other autoimmune diseases, established in the medical history and laboratory findings with positive results for the determination of antinuclear antibodies, anti-cardiolipin antibodies, lupus anticoagulant or direct Coombs test.
7. Patients who are deemed unsuitable for the study by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07; Primary Completion 2013-07 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
Evaluation of platelet response(Chronic ITP) | up to 1 year per subject
  Chronic ITP is defined as having platelet count less than 100×10^9/L,lasting for more than 12 months.
Evaluation of platelet response (Complete Response) | up to 1 year per subject
  CR. A complete response (CR) was defined as a sustained (≥ 3 months) platelet count ≥ 100×10^9/L without recurrence of thrombocytopenia
Evaluation of platelet response (R) | up to 1 year per subject
  R. A response (R) was defined as a sustained (≥ 3 months) platelet count ≥ 30×10^9/L without recurrence of thrombocytopenia

CONTACTS AND LOCATIONS:
Overall Officials: Ming Hou, Dr., Principal Investigator — Shandong University
Locations (1):
- Qilu Hospital, Shandong University, Jinan, Shandong, China

REFERENCES:
- [Result] Medeot M, Zaja F, Vianelli N, Battista M, Baccarani M, Patriarca F, Soldano F, Isola M, De Luca S, Fanin R. Rituximab therapy in adult patients with relapsed or refractory immune thrombocytopenic purpura: long-term follow-up results. Eur J Haematol. 2008 Sep;81(3):165-9. doi: 10.1111/j.1600-0609.2008.01100.x. Epub 2008 May 27. PMID 18510702
- [Result] Provan D, Stasi R, Newland AC, Blanchette VS, Bolton-Maggs P, Bussel JB, Chong BH, Cines DB, Gernsheimer TB, Godeau B, Grainger J, Greer I, Hunt BJ, Imbach PA, Lyons G, McMillan R, Rodeghiero F, Sanz MA, Tarantino M, Watson S, Young J, Kuter DJ. International consensus report on the investigation and management of primary immune thrombocytopenia. Blood. 2010 Jan 14;115(2):168-86. doi: 10.1182/blood-2009-06-225565. Epub 2009 Oct 21. PMID 19846889
- [Result] Rodeghiero F, Stasi R, Gernsheimer T, Michel M, Provan D, Arnold DM, Bussel JB, Cines DB, Chong BH, Cooper N, Godeau B, Lechner K, Mazzucconi MG, McMillan R, Sanz MA, Imbach P, Blanchette V, Kuhne T, Ruggeri M, George JN. Standardization of terminology, definitions and outcome criteria in immune thrombocytopenic purpura of adults and children: report from an international working group. Blood. 2009 Mar 12;113(11):2386-93. doi: 10.1182/blood-2008-07-162503. Epub 2008 Nov 12. PMID 19005182
- [Result] Cheng Y, Wong RS, Soo YO, Chui CH, Lau FY, Chan NP, Wong WS, Cheng G. Initial treatment of immune thrombocytopenic purpura with high-dose dexamethasone. N Engl J Med. 2003 Aug 28;349(9):831-6. doi: 10.1056/NEJMoa030254. PMID 12944568
- [Result] Mazzucconi MG, Fazi P, Bernasconi S, De Rossi G, Leone G, Gugliotta L, Vianelli N, Avvisati G, Rodeghiero F, Amendola A, Baronci C, Carbone C, Quattrin S, Fioritoni G, D'Alfonso G, Mandelli F; Gruppo Italiano Malattie EMatologiche dell'Adulto (GIMEMA) Thrombocytopenia Working Party. Therapy with high-dose dexamethasone (HD-DXM) in previously untreated patients affected by idiopathic thrombocytopenic purpura: a GIMEMA experience. Blood. 2007 Feb 15;109(4):1401-7. doi: 10.1182/blood-2005-12-015222. Epub 2006 Oct 31. PMID 17077333